CLINICAL TRIAL: NCT02164396
Title: Impact of Soft Contact Lenses on Lid-Parallel Conjunctival Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR-005277
Record Dates: First submitted 2013-05-02; First posted 2014-06-16 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-10

CONDITIONS: Lid-Parallel Conjunctival Folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Spectacles Lens (Active Comparator): Participant will discontinue soft contact lens wear and wear spectacles only. Spectacle lens refers to the habitual prescription glasses that the participant arrives to the testing center with; they are NOT prescribed or given to the participant by the investigator as part of the study protocol.
  Interventions: Device: Spectacle Lens
- Habitual Soft Contact Lens (Active Comparator): Participant will continue to wear their habitual soft contact lenses. Habitual lenses are the contact lenses used by the subjects prior to participating in the clinical trial. Various types/brands are used by subjects prior to participation.
  Interventions: Device: Habitual Soft Contact Lens
- Test Lens (Experimental): Participants will be dispensed senofilcon A or narafilcon A depending on their habitual modality (reusable or daily disposable)
  Interventions: Device: Test Lens

INTERVENTIONS:
Device: Spectacle Lens — Spectacle Lens Only
  Arms: Spectacles Lens
Device: Habitual Soft Contact Lens — subject's own contact lens
  Arms: Habitual Soft Contact Lens
Device: Test Lens — senofilcon A or narafilcon A
  Arms: Test Lens

SUMMARY:
The aim of the study is to investigate how Lid-Parallel Conjunctival Folds recovers or persists after the continued usage or discontinuation of contact lenses or refitting with low coefficient of friction lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand and sign the statement of informed consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be 18 years old.
4. The subject's contact lens correction must be in the range of -12.00 to +8.00 in each eye.
5. The subject's refractive cylinder must be less than 1.50D in each eye.
6. The subject must have best visual acuity of 20/40 or better in each eye.
7. The subject must demonstrate adequate mobility and 20/40 vision OD and OS with their habitual contact lenses.
8. The subject must be an adapted soft contact lens wearer in both eyes with at least 1 year experience in contact lens wear.
9. The subject must have normal eyes (i.e. no ocular medications or infections of any type).
10. The subject must have Lid-Parallel Conjunctival Folds greater than or equal to grade 1 OD or OS.

Exclusion Criteria:

1. Currently self reported pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear. This may include, but not be limited to, ocular/systemic pathology or allergy known to affect the conjunctiva, Sjogren's Syndrome, rheumatoid arthritis, diabetes, infections, hay-fever, or if they have had ocular surgery.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
5. Any previous, or planned ocular or intra-ocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
6. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection)on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g. past peripheral ulcer or round peripheral scar), or any other abnormality that may contraindicate contact lens wear.
7. Any ocular infection.
8. Monovision or multi-focal contact lens correction.
9. Participation in any contact lens or lens care product clinical trial within 90 days prior to study enrollment.
10. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV,by self report).
11. Employee of the investigational clinic (e.g. Investigator, Coordinator, Technician)
12. Contact lens wearing of OASYS or TruEye lenses
13. Contact lens wearing time less than 6h/day and/or 5 days/week
14. Extended wear of contact lenses.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weinheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 subjects were enrolled in this study. Of the enrolled subjects all 30 were dispensed study lenses and completed all study visits.
Groups:
- Spectacles: Consists of subjects that were randomized to wear spectacles throughout the duration of the study.
- Habitual Soft Contact Lens: Consists of subjects that were randomized to wear their habitual lens and are the contact lenses used by the subjects prior to participating in the clinical trial. Various types/brands are used by subjects prior to participation.
- Senofilcon A or Narafilcon A: Consists of subjects that were randomized to receive the test lens. In this study there are 2 test lenses. Subjects that were randomized to the test lens were further stratified to either senofilcon A or narafilcon A based on the modality of the habitual contact lens (senofilcon A: Reusable; narafilcon A: Daily Disposable).
Period: Overall Study
Arm/Group | Spectacles | Habitual Soft Contact Lens | Senofilcon A or Narafilcon A
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were randomized to a study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spectacles | Habitual Soft Contact Lens | Senofilcon A or Narafilcon A | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.40 (10.013) | 33.60 (11.918) | 29.0 (9.821) | 32.67 (10.613)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 10 | 25
  Male | 2 | 3 | 0 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Lid-Parallel Conjunctival Folds (LIPCOF)
Description: LIPCOF was assessed at baseline to 2-, 4-, 8- and 12- week Follow-up. Each subject eye was graded using a 4- point using the scale (Grade 0: No conjunctival folds, Grade 1: One permanent and clear parallel fold, Grade 2: Two permanent and clear parallel folds, (normally lower than 0.2mm) and Grade 3: More than two permanent and clear parallel folds, (normally higher than 0.2mm) at two 2 locations in the eye (Temporal and Nasal). The graded responses for each location (Temporal and Nasal) was average. The sum of the average LIPCOF grade for Temporal and Nasal was reported. (Score=average Nasal Grade + average Temporal Grade).
Time Frame: Baseline, 2-, 4-, 8- and 12-Week Follow-up
Population: The analysis population consists of all subjects that completed the study without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: observations
Arm/Group | Spectacles | Habitual Soft Contact Lens | Senofilcon A or Narafilcon A
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (observations) | 20 | 20 | 20
Score
  Baseline | 1.95 (1.050) | 1.75 (1.070) | 1.70 (0.923)
  2-Week Follow-up | 1.40 (1.353) | 2.25 (1.020) | 1.55 (1.276)
  4-Week Follow-up | 1.30 (1.455) | 1.95 (0.826) | 1.05 (1.099)
  8-Week Follow-up | 1.50 (0.946) | 2.15 (1.309) | 1.10 (1.071)
  12- Week Follow-up | 1.35 (0.933) | 2.15 (1.137) | 1.00 (0.795)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 12- weeks per subject.
Arm/Group | Spectacles | Habitual Soft Contact Lens | Senofilcon A or Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days